## **COVER PAGE**

**Title of document:** Randomized Controlled Study of Intraincisional Infiltration Versus Intraperitoneal Instillation of Standardized Dose of Ropivacaine 0.2% in Post-Laparoscopic Cholecystectomy Pain

NCT Number – Not Available

**Document Date** – 01/04/2014

## **Statistical Analysis**

At the end of the study, the envelopes were opened and statistical calculations were made. Mean and standard deviation were observed for continuous forms of data like age, operative duration, numeric pain scores and so on. Such data was further evaluated for significance by Student t-test (for comparing 2 groups), analysis of variance (ANOVA) (for comparing more than 2 groups) and post-hoc analysis in the form of Tukey's Honest Significance Difference (HSD) test. Tukey's HSD test is more conservative in nature as compared to t-test, so has more value in interpretation of results. So, wherever the findings of t-test and Tukey's HSD test disagreed, the results of latter presided over the former. For categorical data, such as results of VDS, FPS-R, ATS and so on, significance testing is done by Fisher's Exact test (FET). A p-value of less than 0.05 was considered statistically significant for all practical applications. Data analysis was done with *IBM SPSS Statistics* \*\* software version 24.